CLINICAL TRIAL: NCT02368158
Title: Reha Drive: Predictors of Fitness to Drive a Car for Cardiologic Patients in Rehabilitation and Acute Clinic and Contactless Determination of Vital Signs Via Camera
Brief Title: Reha Drive: Predictors of Fitness to Drive a Car for Cardiologic Patients and Determination of Vital Signs
Acronym: RehaDrive
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: RWTH Aachen University (Other)
Collaborators: Philips Electronics Nederland B.V. acting through Philips CTO organization (Industry); RWTH Aachen Germany Institut fuer Kraftfahrzeuge (IKA) (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: CTC-A 13-095
Record Dates: First submitted 2015-02-04; First posted 2015-02-20 (Estimated); Last update posted 2015-09-16 (Estimated); Status verified 2015-09

CONDITIONS: Cardiovascular Diseases
Keywords: myocard infarction; arrhythmia; fitness of driving
MeSH Terms: conditions — Cardiovascular Diseases; Arrhythmias, Cardiac

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cardiologic Patient (Experimental): Driving simulation with elevation of medical data in comparison to Lane Change Test plus automotive monitoring via contactless sensors
  Interventions: Other: Driving simulation with elevation of medical data in comparison to Lane Change Test plus automotive monitoring via contactless sensors
- Control Proband (Experimental): The same intervention as in arm "cardiologic patients" :Driving simulation with elevation of medical data in comparison to Lane Change Test plus automotive monitoring via contactless sensors
  Interventions: Other: Driving simulation with elevation of medical data in comparison to Lane Change Test plus automotive monitoring via contactless sensors

INTERVENTIONS:
Other: Driving simulation with elevation of medical data in comparison to Lane Change Test plus automotive monitoring via contactless sensors — During a driving simulation medical data are elevated such as electrocardiography (ECG), heart rate breathing rate and oxygen saturation and compared to data of the performed Lane Change Test as a measurement for the quality of driving. Hereby the deviation of the lane from baseline during driving and ordered lane change via signs are determined also when performing cognitive and visual tasks. Also the simulation is simultaneously accompanied by monitoring via contactless camera usage in regard to possible determination of heart and breathing rate according to Eulerian Magnification Method

SUMMARY:
In this study predictors of fitness to drive a car in cardiologic patients after acute intervention and discharge from hospital to home or rehabilitation are determined in addition to possible automotive monitoring of vital signs via contact less sensors.

DETAILED DESCRIPTION:
Increasing numbers of elderly people with cardiovascular diseases and the wish to drive a car need recommendations corresponding to fitness of driving after their discharge from hospital to home or rehabilitation. A policy paper of the German Cardiac Society (DGK) of 2010 discusses the aptitude of driving a car of cardiovascular patients on experience but only little trial data.Therefore predictors of reduced fitness to drive a car are determined via medical data in comparison to data elevated while "driving" in a simulator and evaluated via Lane Change Test (LCT). Also monitoring of the fitness of driving in the car, automotive monitoring via contactless sensors, could be helpful for judgement.Therefore possible evaluation of heart and breathing rate will be examined with contactless measurements via video camera.

ELIGIBILITY:
Inclusion Criteria:

* cardiologic disease after acute event (e. g. myocard infarction, bypass surgery, device implantation)
* rehabilitation in clinic "An der Rosenquelle"

Exclusion Criteria:

* dementia
* lack of language ability
* pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2013-10; Primary Completion 2015-12 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Electrocardiography (ECG) | 30 minutes
  determination of predictors of fitness of driving a car in cardiologic patients in rehabilitation and acute clinic via comparison of medical data such as ECG, heart rate, breathing rate, oxygen saturation to quality of driving data via Lane Change Test
Breathing rate (BR) | every 5 minutes for 30 minutes
  determination of predictors of fitness of driving a car in cardiologic patients in rehabilitation and acute clinic via comparison of medical data such as ECG, heart rate, breathing rate, oxygen saturation to quality of driving data via Lane Change Test
Heart rate (HR) | every 5 minutes for 30 minutes
  determination of predictors of fitness of driving a car in cardiologic patients in rehabilitation and acute clinic via comparison of medical data such as ECG, heart rate, breathing rate, oxygen saturation to quality of driving data via Lane Change Test
Blood pressure | every 5 minutes for 30 minutes
  determination of predictors of fitness of driving a car in cardiologic patients in rehabilitation and acute clinic via comparison of medical data such as ECG, heart rate, breathing rate, oxygen saturation to quality of driving data via Lane Change Test
oxygen saturation | 30 minutes
  determination of predictors of fitness of driving a car in cardiologic patients in rehabilitation and acute clinic via comparison of medical data such as ECG, heart rate, breathing rate, oxygen saturation to quality of driving data via Lane Change Test
mean deviation of baseline lane | 30 minutes
  determination of predictors of fitness of driving a car in cardiologic patients in rehabilitation and acute clinic via comparison of medical data such as ECG, heart rate, breathing rate, oxygen saturation to quality of driving data via Lane Change Test
mean reaction time | 30 minutes
  determination of predictors of fitness of driving a car in cardiologic patients in rehabilitation and acute clinic via comparison of medical data such as ECG, heart rate, breathing rate, oxygen saturation to quality of driving data via Lane Change Test

SECONDARY OUTCOMES:
heart rate (HR) | every 5 minutes for 30 minutes
  feasibility of automotive monitoring of heart and breathing rate via contactless camera
Breathing rate | every 5 minutes for 30 minutes
  feasibility of automotive monitoring of heart and breathing rate via contactless camera

CONTACTS AND LOCATIONS:
Overall Officials: Sebastian Reith, MD, Principal Investigator — Department of Cardiology, Angiology, Pneumology and Intensive Medicine, RWTH Aachen University Hospital; Skobel Erik, MD, Principal Investigator — Rehabilitation Clinic "Ander Rosenquelle", Kurbrunnenstreet 5, 52066 Aachen
Locations (2):
- Germany (2):
  - Clinic of Rehabilitation "An der Rosenquelle", Aachen, North Rhine-Westphalia
  - Clinic of Cardiology, Angiology, Pneumology and Intensive Medicine, University Hospital Aachen, Aachen, North Rhine-Westphalia